CLINICAL TRIAL: NCT05976074
Title: A Prospective Feasibility Study Evaluating the Use of Wearable Devices to Quantify Tolerance to Deep Brain Stimulation in Essential Tremor Patients
Brief Title: A Study of Wearable Device in Essential Tremor Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bryan T. Klassen, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-004705
Record Dates: First submitted 2023-07-03; First posted 2023-08-04 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Essential Tremor
Keywords: Deep Brain Stimulation Therapy
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Wearable device for tremor assessment (Experimental): Subjects already implanted with a deep brain stimulation (DBS) system for therapy for essential tremor wear an Apple Watch and complete tremor assessment tasks detailed through the BrainRISE app four times a day for two weeks.
  Interventions: Device: Apple Watch; Other: BrainRISE app

INTERVENTIONS:
Device: Apple Watch — The smartwatch will collect data including accelerometry, heart rate, activity, move time, exercise time, stand time, steps, walking and running distance, heart rate variability, respiratory rate, six-minute walk, and flights climbed. During sleep, the smartwatch will collect daily nighttime physiologic data such as time in bed, average sleep time, sleep efficiency, wake after sleep onset, nocturnal heart rate, and nocturnal respiratory rate.
Other: BrainRISE app — The app will play a prerecorded video, which will walk participants through tasks which include holding your arms in different postures, repeating different vowel sounds and phrases as prompted, and tracing different patterns on the phone screen. The tasks are video and audio recorded while being completed. Completing the tremor assessment tasks will take about 10 minutes.

SUMMARY:
The purpose of this research is to observe the daily loss of benefit from DBS therapy by performing a standardized set of tasks throughout the day while wearing an Apple Watch to collect movement and other physiological data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with well-classified essential tremor, who are already receiving regular DBS therapy at Mayo Clinic for their movement disorder.
* Ability to understand study procedures and to comply with them for the entire length of the study and use study devices as outlined in protocol.
* Patient agrees to perform daily tasks in BrainRISE app and consents to the study collecting video and audio recordings during those tasks.
* Proficient in the use of a smart phone.

Exclusion Criteria:

* Cognitive or psychiatric condition rendering a patient unable to cooperate with data collection, or to manage and recharge smart watch and tablet computer devices.
* Presence of open or healing wounds near monitoring sites (infection risk).
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Acquire high-quality physiological signal characteristics from movement disorder patients. | 12 Months
  Acquisition of high-quality physiological signals from 50 subjects with movement disorders over the course of two weeks and up to thirty subjects over one day with 90% compliance rate as determined by the number of study tasks completed by participants.
Acquire high-quality physiological tremor signals from movement disorder patients. | 12 Months
  Measured by wrist accelerometry, which tracks the acceleration of the patients' wrists and is reported in m/sec^2 on a scale where 1.0 = 9.8m/s^2.

SECONDARY OUTCOMES:
Subject feedback | 12 Months
  Subject comfort, compliance, and convenience during the data collection as determined by a post-study assessment asking patients to rate their experience on a scale of 1-5 from hardest and most inconvenient to easiest and least inconvenient.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Klassen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No